CLINICAL TRIAL: NCT01921712
Title: A Phase I, 2-Part, Single-dose, Placebo and Active-Controlled, Dose-ranging, Trial to Evaluate Pharmacokinetics, Pharmacodynamics, Safety and Tolerability in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Safety, Pharmacokinetic and Pharmacodynamic Study of PUR0200 in COPD Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pulmatrix Inc. (Industry)
Collaborators: Quotient Clinical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 601-0010P
Record Dates: First submitted 2013-08-09; First posted 2013-08-13 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- PUR0200 low dose (Experimental): PUR0200 low dose, single dose inhalation
  Interventions: Drug: PUR0200
- PUR0200 mid dose (Experimental): PUR0200 mid dose, single dose inhalation
  Interventions: Drug: PUR0200
- PUR0200 high dose (Experimental): PUR0200 high dose, single dose inhalation
  Interventions: Drug: PUR0200
- Placebo (Placebo Comparator): PUR0200 matched placebo, single dose, inhalation
  Interventions: Drug: PUR0200 Placebo
- Active Comparator (Active Comparator): Active Comparator, single dose, inhalation
  Interventions: Drug: Active comparator

INTERVENTIONS:
Drug: PUR0200 — Randomized single doses of 3 selected doses of PUR0200, compared to a placebo and active comparator
  Arms: PUR0200 high dose; PUR0200 low dose; PUR0200 mid dose
Drug: PUR0200 Placebo — Randomized, single dose of inhaled placebo matched to PUR0200
  Arms: Placebo
Drug: Active comparator — Randomized single dose of inhaled active comparator product
  Arms: Active Comparator

SUMMARY:
The purpose of this study is to assess the safety and tolerability of PUR0200. In addition, the study will look at the blood levels of different doses of PUR0200 and their affect on lung function in COPD patients.

DETAILED DESCRIPTION:
This is a multi-center, 2-part, pharmacokinetic (PK), pharmacodynamic (PD) effect, safety and tolerability study of single doses of PUR0200.

ELIGIBILITY:
Key Inclusion Criteria:

* A clinical diagnosis of moderate to severe COPD according to the following criteria:

  * Current or ex-smokers with at least 10 pack-year smoking history
  * Post-bronchodilator FEV1 >/= 35% and </= 80% of predicted normal value
  * Post-bronchodilator FEV1/FVC (forced vital capacity) ratio <0.70
  * Post-bronchodilator improvement in FEV1 >/= 100 mL

Key Exclusion Criteria:

* Current evidence or recent history of clinically significant or unstable disease (other than COPD)
* Current diagnosis of asthma
* Presence of history of clinically significant allergy requiring treatment
* COPD exacerbation within 6 weeks
* Use of daily oxygen therapy > 10 hours
* Thoracotomy with pulmonary resection
* Use of systemic steroids within 3 months
* Lower respiratory tract infection within 30 days
* Upper respiratory tract infection within 30 days requiring treatment with antibiotics
* History of tuberculosis, bronchiectasis, or other non-specific pulmonary disease
* Prolonged corrected QT (QTc) interval >450 msec males and >470 msec females, or history of long QT syndrome

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) of PUR0200 | 0 to 24 hours
Time to reach peak plasma (Tmax) concentration of PUR0200 | 0 to 24 hours
Area under the plasma concentration versus time (AUC) of PUR0200 | 0 to 24 hours
Trough forced expiratory volume in 1 second (FEV1) | 24 hours
Trough FEV1 difference from baseline | 24 hours
Number of participants with adverse events | up to 14 days post-dose
  adverse events, vital signs, clinical laboratory changes, and ECG changes will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: David Hava, Ph.D., Study Director — Pulmatrix Inc.
Locations (2):
- United Kingdom (2):
  - Medicines Evaluation Unit, Manchester
  - Quotient Clinical, Nottingham